CLINICAL TRIAL: NCT03109535
Title: MapTrek for Sedentary Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Lucas Carr, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201608733
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit-only Group (Active Comparator): Participants received a Fitbit Zip activity monitor to wear daily for 10 weeks.
  Interventions: Behavioral: Fitbit only
- Fitbit + MapTrek Group (Experimental): Participants received a Fitbit Zip activity monitor to wear daily for 10 weeks. Participants also received access to an mHealth game called MapTrek for 10 weeks. MapTrek places users in weekly walking races and sends automated text messages to participants on a daily basis. Messages include a link to the online game as well as motivational messages designed to increase physical activity.
  Interventions: Behavioral: Fitbit + Maptrek

INTERVENTIONS:
Behavioral: Fitbit + Maptrek — Users receive a Fitbit Zip to wear daily. Users aslo receive the mHealth MapTrek game that places users in weekly walking races and sends automated text messages to users on a daily basis for the purpose of increasing daily physical activity.
  Arms: Fitbit + MapTrek Group
Behavioral: Fitbit only — Users receive a Fitbit Zip to wear daily.
  Arms: Fitbit-only Group

SUMMARY:
The aim of this study is to determine if participants randomized to our mHealth MapTrek game increases daily physical activity (average steps/day, active minutes/day) compared to a control group among sedentary office workers over 10 weeks. The investigators hypothesize the MapTrek intervention group will significantly increase their daily steps and active minutes compared to the control group over 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were 21 to 65 year of age, working full-time (at least 35 hours/week) in a desk-dependent job (self-report sitting >75% of work day), who owned a smart phone.

Exclusion Criteria:

* Exclusion criteria included ages <18 years or >65 years, pregnancy or planned pregnancy, prisoner status, and any contraindications to engaging in regular physical activity as identified by the Physical Activity Readiness Questionnaire (PAR-Q), not owning a smart phone, (Cardinal, Esters, & Cardinal, 1996).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Average daily steps | 10 weeks
  Total daily steps as recorded by the Fitbit Zip

SECONDARY OUTCOMES:
Average daily active minutes | 10 weeks
  Minutes with at least 100 steps/minute as recorded by the Fitbit Zip

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gremaud AL, Carr LJ, Simmering JE, Evans NJ, Cremer JF, Segre AM, Polgreen LA, Polgreen PM. Gamifying Accelerometer Use Increases Physical Activity Levels of Sedentary Office Workers. J Am Heart Assoc. 2018 Jul 2;7(13):e007735. doi: 10.1161/JAHA.117.007735. PMID 29967221